CLINICAL TRIAL: NCT04311723
Title: Ventilatory Strategy to Prevent Atelectasis During Bronchoscopy Under General Anesthesia (VESPA Trial)
Brief Title: Ventilatory Strategy for the Prevention of Atelectasis During Bronchoscopy Under General Anesthesia, VESPA Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2019-0387; NCI-2020-00704 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0387 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-03

CONDITIONS: Lung Disorder
MeSH Terms: conditions — Lung Diseases | interventions — Anesthesia; Bronchoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Image reviewers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (conventional mechanical ventilation) (Active Comparator): Patients receive anesthesia using a standard short breathing tube called LMA and then undergo standard of care bronchoscopy.
  Interventions: Procedure: Anesthesia Procedure; Procedure: Bronchoscopy
- Group II (VESPA) (Experimental): Patients receive anesthesia using a longer breathing tube called an endotracheal tube and then undergo standard of care bronchoscopy.
  Interventions: Procedure: Anesthesia Procedure; Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Anesthesia Procedure — Receive anesthesia using laryngeal mask
  Other Names: anesthesia
  Arms: Group I (conventional mechanical ventilation)
Procedure: Anesthesia Procedure — Receive anesthesia using endotracheal tube
  Other Names: anesthesia
  Arms: Group II (VESPA)
Procedure: Bronchoscopy — Undergo standard of care bronchoscopy

SUMMARY:
This trial compares two different types of ventilation for the prevention of partial or complete collapsed lung (atelectasis) in patients undergoing bronchoscopy under general anesthesia. Ventilatory strategy to prevent atelectasis (VESPA) may work better than standard of care mechanical ventilation to reduce the intra-procedural development of atelectasis during bronchoscopy under general anesthesia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if our ventilatory strategy to prevent atelectasis (VESPA) can reduce the intra-procedural development of atelectasis during bronchoscopy under general anesthesia when compared with conventional mechanical ventilation.

SECONDARY OBJECTIVES:

I. To describe proportion of VESPA-induced complications. II. To describe and compare proportion of bronchoscopy-induced complications in VESPA and control arms.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive anesthesia using a standard short breathing tube called laryngeal mask airway (LMA) and then undergo standard of care bronchoscopy.

GROUP II: Patients receive anesthesia using a longer breathing tube called an endotracheal tube and then undergo standard of care bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing bronchoscopy with radial probe endobronchial ultrasound (RP-EBUS) for peripheral lung lesions
* Recent (< 4 weeks) chest computed tomography (CT) performed prior to the bronchoscopy
* Voluntary informed consent to participate in the study

Exclusion Criteria:

* Patients with baseline lung consolidation, interstitial changes or lung masses (> 3 cm in diameter) in dependent areas of the lung (right/left [R/L] B6, 9, or 10 bronchial segments) as seen on most recent CT
* Pregnancy
* Ascites
* Known diaphragmatic paralysis
* Air-trapping with residual volume > 150% of predicted
* History of primary or secondary spontaneous pneumothorax
* Lung bullae > 5 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Presence or absence of new atelectasis for each segment | At the time of bronchoscopy
  The proportion of patients identified as developing intraprocedural atelectasis by radial probe endobronchial ultrasound (RP-EBUS) and its 95% confidence interval will be estimated. The proportion of patients developing intraprocedural atelectasis will be compared between treatment and control arms, utilizing a 2-sided Chi-square test or Fisher's exact test to accomplish primary objective. Locations of atelectasis will be summarized in a frequency table, allowing for multiple locations in the same patient. The proportion of segments identified as developing atelectasis among all evaluated segments will be calculated for each patient, and the distribution of the proportion will be summarized by the mean, median, and range.
Presence or absence of atelectasis within each of the 6 bronchial segments | During preoperative computed tomography (CT)
  Will be determined using RP-EBUS. A segment will be identified as having a new atelectasis if there is an indication of solid- or semisolid-appearing lesion by RP-EBUS without a corresponding indication of solid tumor or atelectasis on the preoperative CT. If any of the two subsegments of any specific center has atelectasis, that segment will be considered atelectatic. The outcome of the reading will be defined by whatever pattern 2 or all 3 readers agree on. Locations of atelectasis will be summarized in a frequency table, allowing for multiple locations in the same patient. The proportion of segments identified as developing atelectasis among all evaluated segments will be calculated for each patient, and the distribution of the proportion will be summarized by the mean, median, and range.
Presence or absence of atelectasis for each patient | Up to 1 year
  After identifying the presence or absence of new atelectasis for each segment, patients with at least 1 segment containing a new atelectasis will be determined to have atelectasis. Patients without atelectasis in any of the 6 segments will be determined to not have atelectasis. Patients with atelectasis and patients without atelectasis will be compared in terms of patient characteristics using a t-test or Wilcoxon test for continuous variables and Fisher's exact test or Chi-squared test for categorical variables.

SECONDARY OUTCOMES:
Ventilatory strategy to prevent atelectasis (VESPA)-induced complications | Within 48 hours of bronchoscopy
  Proportion of VESPA-induced complications will be estimated along with 95% credible interval.
Bronchoscopy-induced complications | Within 48 hours of bronchoscopy
  Proportion of bronchoscopy-induced complications between VESPA and control arms will be estimated and compared by Chi-square test or Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto F Casal, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Salahuddin M, Sarkiss M, Sagar AS, Vlahos I, Chang CH, Shah A, Sabath BF, Lin J, Song J, Moon T, Norman PH, Eapen GA, Grosu HB, Ost DE, Jimenez CA, Chintalapani G, Casal RF. Ventilatory Strategy to Prevent Atelectasis During Bronchoscopy Under General Anesthesia: A Multicenter Randomized Controlled Trial (Ventilatory Strategy to Prevent Atelectasis -VESPA- Trial). Chest. 2022 Dec;162(6):1393-1401. doi: 10.1016/j.chest.2022.06.045. Epub 2022 Jul 6. PMID 35803302
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT04311723/ICF_000.pdf